CLINICAL TRIAL: NCT03006484
Title: Neurological Outcomes After In-hospital Cardiac Arrest: a Prospective Observational Study
Brief Title: Neurological Outcomes After In-Hospital Cardiac Arrest
Acronym: NO-IHCA
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sang-Beom Jeon, Associate Professor, Asan Medical Center
Other Study IDs: 2016-1378
Record Dates: First submitted 2016-12-26; First posted 2016-12-30 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Inhospital Cardiac Arrest
Keywords: Cardiac arrest; Inhospital Cardiac Arrest; Cardiopulmonary Resuscitation
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Before Period: Patients who developed in-hosptial cardiac arrest before the implementation of new legislation on life-sustaining treatments
- After Period: Patients who developed in-hosptial cardiac arrest after the implementation of new legislation on life-sustaining treatments
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will be needed.
  Groups: After Period

SUMMARY:
Little is known about the long-term neurological outcomes after in-hospital cardiac arrest (IHCA). It is also not known whether withdrawal of life-sustaining measures will influence rates of survivors with poor neurological status. Currently, withdrawal of care in comatose patients after cardiac arrest is strongly forbidden by law in Korea. However, a new legislation on allowing withdrawal of care will come into effect since early 2018 in Korea. The investigators aim to determine 1) long-term neurological outcomes in patients who developed IHCA, 2) whether early neurological status can predict late neurological status after IHCA, and 3) whether the proportion of IHCA survivors with good neurological outcomes will change since implementation of new legislation on withdrawal of care.

DETAILED DESCRIPTION:
<The schedule of assessment>

* Day 0: Neurological examination (First examination will be performed within 2 hours after IHCA)
* Day1 - 7: Neurological examination
* Day7, 14, 21, 28: Neurological examination, CPC score
* Day90: CPC score, survival
* Day180: CPC score, survival
* Day 360: CPC score, survival

<Cerebral Performance Category(CPC) score>

* CPC 1: good cerebral performance
* CPC 2: Moderate cerebral disability(available for independent activities)
* CPC 3: Severe cerebral disability(dependent on others for daily support)
* CPC 4: Coma or vegetative state
* CPC 5: Brain death or death

<Acronyms>

* ACDU(Alert/Confused/Drowsy/Unresponsive) score
* FOUR(Full Outline of Unresponsiveness) score

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* In-hospital cardiac arrest
* Cardiopulmonary Resuscitation(CPR) code activation and/or neurology consultation for IHCA

Exclusion Criteria:

* Neither (CPR) code activation nor neurology consultation
* Development of IHCA during transition period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient who experienced In-hospital cardiac arrest(IHCA) in Asan Medical Center.
Sampling Method: Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
Cerebral Performance Category(CPC) score of 1-2 | 12 month after In-Hospital Cardiac Arrest(IHCA)
  CPC score is the most universal index to assess neurological outcome following cardiac arrest. CPC score is classified according to the point. Good neurological outcome is defined as CPC 1-2 and poor is CPC 3-5.
  CPC score will be evaluated by neurological examination and the results of other exam.
  * Neurological examination: Neurologist will perform directly until the point of CPC score 1 is confirmed.
    1. mental status: ACDU score, FOUR score and Glasgow Coma Scale
    2. brain stem reflex: Light reflexes by pupillometer(the NeurOptics® NPi™-100 (Neuroptics Inc., Irvine, CA, USA)) and corneal reflexes
    3. motor status
       * Responsive state: Medical Research Council grade
       * Unresponsive state: motor response to painful stimuli)
    4. seizure evaluation: status myoclonus , seizure, status epilepticus
  * The result of other examinations in accordance with medical treatment guideline will be evaluated as well. (e.g. Finding MRI of the brain, EEG, neuron specific enolase)

SECONDARY OUTCOMES:
CPC score | Day 7, day 14, day 21, day 28, 3 month, 6 month, and 12 month after IHCA
  CPC score is the most universal index to assess neurological outcome following cardiac arrest. CPC score is classified according to the point. Good neurological outcome is defined as CPC 1-2 and poor is CPC 3-5.
  CPC score will be evaluated by neurological examination and the results of other exam.
  * Neurological examination: Neurologist will perform directly until the point of CPC score 1 is confirmed.
    1. mental status: ACDU score, FOUR score and Glasgow Coma Scale
    2. brain stem reflex: Light reflexes by pupillometer(the NeurOptics® NPi™-100 (Neuroptics Inc., Irvine, CA, USA)) and corneal reflexes
    3. motor status
       * Responsive state: Medical Research Council grade
       * Unresponsive state: motor response to painful stimuli)
    4. seizure evaluation: status myoclonus , seizure, status epilepticus
  * The result of other examinations in accordance with medical treatment guideline will be evaluated as well. (e.g. Finding MRI of the brain, EEG, neuron specific enolase)
Mortality | Day 0-28, 3 month, 6 month, and 12 month after IHCA
  A measure of the number of deaths in a particular population
Awakening | Day 0-28 after IHCA
  Following commands
Neurological recovery | Day 0-28 after IHCA
  CPC of 1

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Beom Jeon, Master, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: No